CLINICAL TRIAL: NCT07308522
Title: Clinical ,Microbiological and Compliance Outcomes of AI-based vs Standard Electric and Manual Toothbrushes in Adults With Plaque-Induced Gingivitis: A 6-Week Randomized Controlled Trial
Brief Title: Clinical ,Microbiological and Compliance Outcomes of AI-based Toothbrushes in Plaque Induced Gingivitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Buthaina Firas Faisal, Researcher, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1120625
Record Dates: First submitted 2025-12-13; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-11

CONDITIONS: Plaque Induced Gingivitis; Toothbrushing; Compliance
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Manual toothbrush (Active Comparator)
  Interventions: Device: Manual toothbrush
- Electric toothbrush (Active Comparator)
  Interventions: Device: Electric toothbrush
- AI-based toothbrush (Experimental)
  Interventions: Device: AI toothbrush

INTERVENTIONS:
Device: AI toothbrush — Smart toothbrush supported with AI applications to improve toothbrushing experience
  Arms: AI-based toothbrush
Device: Manual toothbrush — Manual toothbrush used as a gold standard control
  Arms: Manual toothbrush
Device: Electric toothbrush — Electric toothbrush as a second control group
  Arms: Electric toothbrush

SUMMARY:
Severe periodontitis is widespread and begins with reversible gingivitis, driven by poor oral hygiene and a dysbiotic microbiome. Daily toothbrushing is the simplest prevention, but patients still leave plaque. Electric brushes remove more plaque and reduce gingivitis better than manual ones, and users show better periodontal status. App-connected smart brushes and apps aim to improve adherence. Trials increased plaque reduction and brushing time versus manual brushing, but app layers have not clearly beaten standard power brushes, and microbiological outcomes are rarely reported. Xiaomi's AI-based sonic T501 adds pressure sensing, personalised coaching and coverage tracking, whereas the T302 is a simpler non-connected sonic brush. Streptococcus sanguinis is a health-associated early coloniser; its qPCR-measured relative abundance marks a healthy supragingival profile. It is still unclear whether AI guidance adds extra benefit beyond a standard electric brush in adult gingivitis.

DETAILED DESCRIPTION:
Worldwide, 538 million people are reported to have severe periodontitis .The root of this problem lies in its initial stage, gingivitis. Gingivitis typically results from inadequate oral hygiene, which can quickly shift a healthy oral microbiome to a dysbiotic state, leading to gingival inflammation and bleeding. If this early stage is not treated, more advanced periodontal disease can occur with irreversible oral health consequences and systemic implications.

Among the simplest and most cost-effective approaches for preventing periodontal disease is daily self-care. Effective toothbrushing mechanically removes plaque, reverses gingivitis, and prevents its inception.The better plaque is controlled, the more substantial the clinical gains. However, even with their best efforts, patients often leave considerable amounts of plaque behind after toothbrushing .

Various toothbrush designs and technologies have been developed to improve plaque removal. Results of systematic reviews and meta-analyses evaluating these options consistently showed electric toothbrushes provide significantly greater plaque removal and gingivitis control than manual toothbrushes. These benefits have been corroborated by the results of population-based research showing poorer periodontal health status and fewer teeth present for manual toothbrush users than electric toothbrush users. AI in dentistry uses machine-learning tools to assist clinicians detecting disease on radiographs, supporting diagnosis/risk assessment (e.g., caries/periodontitis), optimizing treatment planning/CAD-CAM, and boosting patient adherence via smart, sensor-based brushes and apps. In early app-connected trials, adolescents used a manual brush and an interactive, Bluetooth-enabled oscillating-rotating brush + app. The app-connected brush significantly increased whole-mouth plaque reduction and brushing time in a 2-week single-blind RCT .

Another was a three-arm, eight-week RCT that compared a manual brush to the same power brush with or without app assistance in dental students with gingivitis.

For plaque and bleeding, both powered brushes performed better than the manual; however, in that sample, the app layer did not provide a definite clinical advantage over the non-app powered brush . Recently, a smart sonic toothbrush (Xiaomi T501) has been introduced that combines a magnetic-levitation motor with motion/pressure sensing and app-based coaching. The motor generates high-frequency micro-vibrations that transmit energy to the bristle tips while the built-in pressure sensor limits excessive force.

Through Bluetooth, the brush can provide real-time timers, quadrant pacing, and zone-coverage feedback in the Xiaomi Home app. In addition, an AI-adjustment module analyzes inertial-sensor and pressure data from prior sessions to personalize guidance, highlighting under-cleaned zones, recommending softer intensity after repeated over-pressure events. Standard electric brush (Xiaomi T302) a non-connected sonic toothbrush with a low-noise brushless motor and 4 cleaning modes. It includes a built-in 2-minute timer with 30-second pacing to cue quadrant changes. The device has no Bluetooth/app (no AI guidance) and no pressure-sensor. Microbiologically, in periodontal health, supragingival plaque is dominated by early colonizing streptococci (e.g., Streptococcus sanguinis, S. mitis, S. gordonii) that form part of the health-associated "yellow/green" groups .

With plaque accumulation , communities follow a reproducible succession:

biomass increases and the microbiota shifts toward more anaerobic, proteolytic taxa (e.g., Fusobacterium, Prevotella), paralleling clinical inflammation . Streptococcus sanguinis is a key health-associated commensal and early enamel colonizer; its presence correlates with clinically healthy plaque and caries- resistance. During gingivitis development, S. sanguinis often decreases as more anaerobic species expand, so we will quantify its relative abundance by qPCR as a marker of a health-associated supragingival profile, reported alongside clinical indices. Evidence gap : Existing app-connected toothbrush trials are mostly comparing powered+app to manual brushing, so they do not isolate whether modern AI-based guidance adds benefit beyond a standard electric brush in adult gingivitis patients . Microbiological endpoints reported in parallel with clinical outcomes are rarely included.

ELIGIBILITY:
Inclusion Criteria:

* Participants should be systemically healthy
* 18 years old, with the presence of ≥ 20 teeth
* Diagnosed with generalized plaque-induced gingivitis having >30% bleeding sites, with probing depths ≤3 mm and intact periodontium
* Participants with at least secondary school education, who are able to read and understand basic English to follow the app-based toothbrush instructions

Exclusion Criteria:

* Participants who using antibiotics or anti-inflammatory medication throughout the investigation or during the previous 3 months prior to the study.
* Drug-induced gingival enlargement (phenytoin, cyclosporine, calciumchannel blockers).
* Individuals with periodontitis and healthy periodontium.
* Mouth breathers .
* Individuals with severe dental crowding or malalignment that prevents proper toothbrushing.
* Individuals with heavy calculus.
* Individuals who smoke or alcoholism.
* Pregnant, breastfeeding women or those using contraceptive tablets.
* Individuals with orthodontic devices or removable dentures

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Plaque index | This index will be recorded at baseline, after 2 weeks, and 2 months after enrollment
  Turesky-modified Quigley-Hein Plaque Index will be quantified on a scale between 0 to 5:
  0 No plaque
  1. Isolated areas of plaque at the cervical margin of the tooth.
  2. A thin continuous band of plaque (up to 1 mm) at cervical margin of tooth.
  3. A band of plaque wider than 1 mm but covering less than one- third of the crown of the tooth.
  4. Plaque covering at least one-third but less than two-thirds of the crown of the tooth.
  5. plaque covering two-thirds or more of the crown of the tooth.

SECONDARY OUTCOMES:
Modified sulcular bleeding index | The index will be recorded at baseline, 2 weeks, and 2 months after enrolment
  Bleeding after probing gingival sulcus will be scored as follows:
  Score 0: No bleeding. Score 1: Isolated spots bleeding. Score 2: Blood forms a confluent red line or margin. Score 3: Heavy or profuse bleeding
Compliance to oral hygiene instructions and level of satisfaction | The compliance will be assessed after 2 week and 2 months. Satisfaction will be assessed at the endpoint of the study (2 months)
  Degree of compliance and patient-reported outcome about satisfaction level after using different types of toothbrushes using a questionnaire
Microbiological analysis | Plaque samples will be collected for analysis at baseline, 2 weeks, and 2 months
  Relative abundance of Streptococcus Sanguinis in supragingival plaque samples will be measured using PCR technique.

CONTACTS AND LOCATIONS:
Locations (1):
- College of Dentistry, University of Baghdad, Baghdad, Al-Rasafa, Iraq

IPD SHARING:
Plan to Share IPD: Yes
Only IPD relevant to study results will be shared. Other personal information such as full names, phone number, location, marital status, and income level will not be shared for confidentiality reasons.